CLINICAL TRIAL: NCT03293264
Title: Effects of a Workplace Health Service Program in Employees With Diagnosed Metabolic Syndrome
Brief Title: Exercise Training on Metabolic Syndrome Severity in Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Volkswagen AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RebVW
Record Dates: First submitted 2017-09-15; First posted 2017-09-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2023-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; exercise training; employees; workplace; operational health service
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise training group (Experimental): The intervention group will be encouraged to perform 150 min of exercise training per week for 6 months. Subjects will be provided with individual feedback and exercise Training prescriptions. After month 6 subjects will be randomized to three different groups for follow-up observation.
  Interventions: Behavioral: Exercise training group
- Waiting-control group (No Intervention): The control group will be provided with general informations on a healthy lifestyle. After 6 months wait-list-control months subjects will receive the guided exercise training intervention for 6 months.

INTERVENTIONS:
Behavioral: Exercise training group — Exercise training will consist of 3 - 6 sessions per week and will cumulate in 150 min net exercise time per week. Heart rates during exercise sessions will be monitored with the aim of physical activities at moderate-intensity. Exercises will be individualized to reach the best possible improvements to the cardiovascular and musculoskeletal system. Possible disciples will include but are not limited to: cycling, rowing (ergometer), swimming, walking, nordic-walking, running, arm-cycle-ergometer or cross-trainer as well as fitness courses offered from occupational or private providers. Everyday activities which reach an effective heart rate range can account for exercise training on a home-based basis .
  Advise on complementary individual strength and coordination exercises will be added to the training program. A nutrition analyses will be completed by every subject to account for special needs of the metabolic syndrome.
  Arms: Exercise training group

SUMMARY:
Hypothesis: An occupational 6 months physical exercise training will lead to better health behaviour and improve the severity of the metabolic syndrome.

312 subjects will be assigned to either an intervention or a waiting-control-group. The intervention group will receive instructions with the aim to perform 150 min exercise training per week. Exercise consists of endurance, strength and coordination training. A feedback system guided by sports scientists will be installed for all subjects in the intervention group using activity monitoring (wearable). After 6 months training subjects from the intervention group will be assigned to one of the following groups for follow-up observation from month 6 to months 12:

* training with personal/individual feedback from sport scientist
* training with automated feedback using activity monitoring Tools (wearable)
* training without further feedback Subjects assigned to the control group will be provided with information on low intensity motion exercises. After 6 months in the control group subjects will be provided with the same exercise intervention as the intervention for a duration of 6 months.

Study visits will be conducted at month 0, month 6, month 12, and a long-term follow-up at month 24..

ELIGIBILITY:
Inclusion Criteria:

* 3 out of 5 parameters of the metabolic syndrome

Exclusion Criteria:

* ongoing participation in occupational health service
* clinical relevant acute or chronic infections
* pregnancy
* surgery dating back less than 8 weeks
* artificial joint replacement dating back less than 6 months
* tumor disease dating back less than 5 years
* every other disease or relevant functional disorder not allowing to participate in regular physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Metabolic Syndrome (MetS) -Z-score | 6 months 12 months, 24 months
  Z-Score (arbitrary unit, ranging from -2 to 2), assessed and calculated from the 5 established components of the metabolic syndrome: triglycerides, HDL cholesterol, fasting glucose, waist circumference, and systolic blood pressure.

SECONDARY OUTCOMES:
Change from baseline in Work-Ability-Index (WAI) | 6 months, 12 months, 24 months
  score of WAI questionnaire, (Outcome work ability score: Minimum 1 Point, Maximum 49 Points)
Change from baseline in Health-related quality of live: score of SF36 questionnaire | 6 months, 12 months, 24 months
  score of SF36 questionnaire (outcomes: physical component score: Minimum 1 Point, Maximum 100 Points, mental component score: Minimum 1 Point, Maximum 100 Points)
Change from baseline in Pmax | 6 months
  Maximum workload reached in an graded exercise test (watt/kg Body Weight).
Change from baseline in Body weight | 6 months
  kg
Change from baseline in body composition | 6 months, 12 months, 24 months
  fat mass (kg), fat free mass (kg), visceral fat mass (kg)
Change from baseline in adherence to training program | 6 months, 12 months, 24 months
  percentage (%) of time (150 min per week) spend on exercising (minutes)
Change from baseline in Anxiety- and depression severity | 6 months, 12 months, 24 months
  Hospital Anxiety and Depression Scale, (outcomes: amxiety severity: Minimum 1 Point, Maximum 21 Points, Depression severity: Minimum 1 Point, Maximum 21 Points)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haverich, Prof. Dr., Study Chair — Hannover Medical School, Department of Cardiothoracic, Transplantation and Vascular Surgery (HTTG); Uwe Tegtbur, Prof. Dr., Study Chair — Hannover Medical School, Institute for Sports Medicine
Locations (1):
- HannoverMS, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayerle P, Haufe S, Kuck M, Protte G, Kerling A, Ewers S, Boeck HT, Sundermeier T, Ensslen R, Kahl KG, Haverich A, Tegtbur U, Nachbar L. The Impact of Body Weight Changes versus Exercise Capacity Changes on Health-Related Factors following a Lifestyle Intervention in Employees with Metabolic Syndrome. Nutrients. 2022 Oct 29;14(21):4560. doi: 10.3390/nu14214560. PMID 36364823
- [Background] Bayerle P, Kerling A, Kuck M, Rolff S, Boeck HT, Sundermeier T, Ensslen R, Tegtbur U, Lauenstein D, Bothig D, Bara C, Hanke A, Terkamp C, Haverich A, Stiesch M, de Zwaan M, Haufe S, Nachbar L. Effectiveness of wearable devices as a support strategy for maintaining physical activity after a structured exercise intervention for employees with metabolic syndrome: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Feb 10;14(1):24. doi: 10.1186/s13102-022-00409-1. PMID 35144658
- [Background] Haufe S, Hupa-Breier KL, Bayerle P, Boeck HT, Rolff S, Sundermeier T, Kerling A, Eigendorf J, Kuck M, Hanke AA, Ensslen R, Nachbar L, Lauenstein D, Bothig D, Hilfiker-Kleiner D, Stiesch M, Terkamp C, Wedemeyer H, Haverich A, Tegtbur U. Telemonitoring-Supported Exercise Training in Employees With Metabolic Syndrome Improves Liver Inflammation and Fibrosis. Clin Transl Gastroenterol. 2021 Jun 18;12(6):e00371. doi: 10.14309/ctg.0000000000000371. PMID 34140456
- [Background] Haufe S, Kahl KG, Kerling A, Protte G, Bayerle P, Stenner HT, Rolff S, Sundermeier T, Eigendorf J, Kuck M, Hanke AA, Keller-Varady K, Ensslen R, Nachbar L, Lauenstein D, Bothig D, Terkamp C, Stiesch M, Hilfiker-Kleiner D, Haverich A, Tegtbur U. Employers With Metabolic Syndrome and Increased Depression/Anxiety Severity Profit Most From Structured Exercise Intervention for Work Ability and Quality of Life. Front Psychiatry. 2020 Jun 18;11:562. doi: 10.3389/fpsyt.2020.00562. eCollection 2020. PMID 32625123
- [Background] Haufe S, Kerling A, Protte G, Bayerle P, Stenner HT, Rolff S, Sundermeier T, Kuck M, Ensslen R, Nachbar L, Lauenstein D, Bothig D, Bara C, Hanke AA, Terkamp C, Stiesch M, Hilfiker-Kleiner D, Haverich A, Tegtbur U. Telemonitoring-supported exercise training, metabolic syndrome severity, and work ability in company employees: a randomised controlled trial. Lancet Public Health. 2019 Jul;4(7):e343-e352. doi: 10.1016/S2468-2667(19)30075-1. Epub 2019 Jun 13. PMID 31204284